CLINICAL TRIAL: NCT00304252
Title: A Phase II, Multicenter, Randomised, Double-blind, Placebo Controlled, Dose Finding Study of Subcutaneously Administered Interferon Beta-1a for Maintenance of Remission in Patients With Crohn's Disease
Brief Title: Safety and Efficacy of Treatment With Interferon Beta-1a Rebif® in Patients With Crohn's Disease
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of Efficacy
Sponsor: EMD Serono (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 22916; 9903
Record Dates: First submitted 2006-03-14; First posted 2006-03-17 (Estimated); Last update posted 2013-08-06 (Estimated); Status verified 2013-08

CONDITIONS: Crohn's Disease
MeSH Terms: conditions — Crohn Disease | interventions — Interferon beta-1a

INTERVENTIONS:
Drug: Interferon beta-1a

SUMMARY:
The purpose of this study is to determine the safety and efficacy of interferon beta-1a in maintaining remission in patients with Crohn's disease.

ELIGIBILITY:
Inclusion Criteria:

* Patients with an established diagnosis of Crohn's disease who went into remission using corticosteroids within 4 weeks before the study

Exclusion Criteria:

* Any other treatment for the maintenance of remission of Crohn's disease

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 192
Dates: Start 2001-11; Study Completion 2003-09 (Actual)

PRIMARY OUTCOMES:
The primary efficacy endpoint was the proportion of patients who maintained remission (relapse-free) and did not receive any additional treatment for the management of Crohn's disease by week 26.

SECONDARY OUTCOMES:
The secondary efficacy endpoints assessed the effect of treatment with IFN beta 1a on the following measures:
The proportion of patients who maintained remission (relapse-free) and did not receive any additional treatment for the management of Crohn's disease by week 52
Time to relapse
Change from baseline to end of treatment in Quality of Life (IBDQ) score, CDAI score, biological markers of inflammation (CRP and ESR), number of fistulas (including new fistulas and closure of existing ones), and antibodies to interferon beta-1a.

CONTACTS AND LOCATIONS:
Overall Officials: Claudia Pena Rossi, M.D., Study Director — EMD Serono
Locations (5):
- Medical Information Office, Munich, Germany
- Medical Information Office, Roma, Italy
- Medical Information Office, Solna, Sweden
- Medical Information Office, Zug, Switzerland
- Medical Information Office, Feltham, United Kingdom

REFERENCES:
- [Derived] Pena Rossi C, Hanauer SB, Tomasevic R, Hunter JO, Shafran I, Graffner H. Interferon beta-1a for the maintenance of remission in patients with Crohn's disease: results of a phase II dose-finding study. BMC Gastroenterol. 2009 Mar 20;9:22. doi: 10.1186/1471-230X-9-22. PMID 19302707
- See also: Full FDA approved prescribing information can be found here — http://www.mslifelines.com